CLINICAL TRIAL: NCT02480192
Title: Cognitive Behavioural Therapy for Menopausal Symptoms: A Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy for Menopausal Symptoms
Acronym: CBTMENO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Sheryl Green, Clinical Health Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMHF-SG1
Record Dates: First submitted 2015-05-22; First posted 2015-06-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Menopausal Depression
Keywords: Vasomotor; Symptoms

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized controlled trial was conducted to assess the effectiveness of the CBT-Meno program compared to a waitlist comparison condition.
Who Masked: Outcomes Assessor
Masking Description: Assessors evaluated symptoms at baseline, 12-weeks post-baseline, and 3-month follow-up. Assessors were unaware of participants' assigned condition.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (CBT-Meno) (Experimental): After an initial assessment, the experimental group received 12 weekly sessions (2 hours each) of group-based cognitive-behavioural therapy for menopausal symptoms (CBT-Meno) (up to n=8 per group). Symptoms that were targeted included vasomotor symptoms (hot flashes/night sweats), depressive symptoms, anxiety, poor sleep, and sexual concerns. Participants were re-assessed at 12-weeks post-baseline and at 3 months post-treatment.
  Interventions: Other: CBT for Menopausal Symptoms (CBT-Meno)
- Waitlist (No Intervention): After an initial assessment, the waitlist comparison group did not receive any treatment for 12 weeks. They were then re-assessed at 12-weeks post-baseline and this data was used to compare this group to the experimental group to determine the effectiveness of the CBT-Meno treatment. After this re-assessment participants in the waitlist condition were offered the same CBT-Meno treatment as the experimental group: 12 weekly sessions (2 hours long) of cognitive-behavioural therapy for menopausal symptoms.

INTERVENTIONS:
Other: CBT for Menopausal Symptoms (CBT-Meno) — This 12-week CBT-based group treatment program consists of a combination of components including: a) psychoeducation about the nature of menopause including examination about thoughts and beliefs, b) cognitive and behavioural modification related to vasomotor symptoms, c) cognitive-behavioural strategies for depression, e) cognitive-behavioural strategies for anxiety and panic, d) sleep hygiene and cognitive-behavioural strategies for sleep difficulties, f) psychoeducation and lifestyle and behavioural modifications for urogenital complaints, and g) psychoeducation and cognitive-behavioural strategies for sexual concerns.
  Arms: Experimental Group (CBT-Meno)

SUMMARY:
This study examined the effectiveness of a new cognitive-behavioural therapy for menopausal symptoms (CBT-Meno). Half of participants were randomly assigned to the 12-week CBT-Meno program and half to a 12-week waitlist. Common menopause symptoms (i.e., hot flashes/night sweats, depression, anxiety, poor sleep, and sexual concerns) were assessed at baseline, 12-weeks post-baseline, and (for women in the CBT-Meno condition) at 3-month follow-up.

DETAILED DESCRIPTION:
Women going through the menopausal transition often experience adverse physical changes (e.g., hot flashes/night sweats, sleep difficulties, sexual concerns) in addition to emotional difficulties (e.g., depression, anxiety) that can significantly impact functioning and overall quality of life. To date, hormone therapy (HT) has been the most commonly used treatment to relieve symptoms of menopause. However, reports have questioned the safety of HT long-term (e.g., risk of heart attacks, strokes, cancer) for some women. Cognitive-behavioural therapy (CBT), has been proposed as a low-risk treatment for menopausal symptoms. The investigators developed a comprehensive non-pharmacological, CBT for menopausal symptoms (CBT-Meno), published the treatment manual (Green, McCabe, & Soares, 2012), and obtained initial evidence supporting the effectiveness of CBT-Meno in a single-sample pilot study (Green et al., 2013). The goal in the study reported here was to conduct a larger randomized controlled trial to evaluate the effectiveness of the CBT-Meno program compared to a waitlist condition. The investigators hypothesized that participants would experience less intense/disruptive hot flashes/night sweats, reduced depression and anxiety, improvement in sleep difficulties, and sexual concerns. The investigators also predicted that these benefits would be maintained at 3-month follow-up and that participants would report high treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal staging: perimenopause or postmenopausal as per STRAW definitions (Harlow et al., 2012) or having surgically-induced menopause
2. A minimum of mild level of severity of depressive symptoms (defined by the Beck Depression Inventory, scores of 14 or greater during initial screen),
3. Significant vasomotor symptoms: i.e., vasomotor symptoms that are (a) frequent (≥ 4 hot flashes per day/night or 21 or more per week); (b) distressing (≥ 3 or more on the vasomotor subscale of the Greene Climacteric Scale); and (c) interfering (≥ 30 or greater on the Hot Flash Related Daily Interference Scale).
4. Not taking hormonal, anti-depressant, or any herbal therapies or if taking these medications they must be taking a stable dose for at least three months prior to the study and for the duration of the study,
5. Speak, read, and write in English sufficiently to comprehend testing procedures and written materials in group treatment.

Exclusion Criteria:

1. Participants who are severely depressed/suicidal at the time of the screen or intake assessment that would warrant acute treatment and hence, render them unable to act as a wait list control participant if randomized to this condition,
2. Participants with Psychotic Disorders, or current Substance Dependence.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The Hot Flash Related Daily Interference Scale | 12 weeks
  The Hot Flash Related Daily Interference Scale assesses the degree to which vasomotor functions interfere with daily life (Carpenter, 2001). The current study aims to explore whether CBGT for menopausal symptoms significantly reduces vasomotor function daily interference, as captured by the Hot Flash Related Daily Interference Scale, compared to pre-treatment and wait-list controls.
The Beck Depression Inventory | 12 weeks
  The Beck Depression Inventory is a multiple choice questionnaire which measures depressive symptoms (Beck, Steer & Brown, 1996). The current study aims to explore whether CBGT for menopausal symptoms significantly reduces subjective depressive symptoms, compared to pre-treatment and wait-list controls.

SECONDARY OUTCOMES:
The Greene Climacteric Scale - Vasomotor Subscale | 12 weeks
  The Greene Climacteric Scale is a self-report questionnaire which measures four menopause-related domains: Vasomotor symptoms, depression and anxiety, physical complaints, and sexual concerns (Greene, 1998). The current study aims to explore whether CBGT for menopausal symptoms significantly improves typical menopausal symptoms, as captured by the Greene Climacteric Scale, compared to pre-treatment and wait list controls?
The Montgomery-Asberg Depression Rating Scale | 12 weeks
  The Montgomery-Asberg Depression Rating Scale (Montgomery & Asberg, 1979) is a measure that requires an interview format assessing depressive symptoms in menopausal women and contains a global severity score. The current study aims to explore whether CBGT for menopausal symptoms significantly reduces menopausal depressive symptoms, as captured by the Montgomery-Asberg Depression Rating Scale, compared to pre-treatment and wait-list controls.
The Hamilton Anxiety Scale | 12 weeks
  The Hamilton Anxiety Scale is an interview format rating scale developed to quantify the severity of anxiety symptomatology and contains a global score (Hamilton, 1956). The current study aims to explore whether CBGT for menopausal symptoms significantly improves objective anxiety symptoms, as captured by the Hamilton Anxiety Scale, compared to pre-treatment and wait list controls.
The Pittsburgh Sleep Quality Inventory | 12 weeks
  The Pittsburgh Sleep Quality Inventory (Buysee et al, 1989) is a self-report inventory that contains seven component scores along with one global score indicating overall sleep quality. The current study aims to explore whether CBGT for menopausal symptoms significantly improves sleep disruption, as captured by the Pittsburgh Sleep Quality Inventory, compared to pre-treatment and wait list controls.
Ambulatory Sternal Skin-Conductance Monitoring | 12 weeks
  Vasomotor symptoms will be assessed objectively through ambulatory sternal skin-conductance monitoring which will be worn for 2 consecutive days prior to each assessment. The current study aims to explore whether CBGT for menopausal symptoms significantly reduces vasomotor symptoms (hot flashes/night sweats) compared to pre-treatment and wait-list controls.
Female Sexual Functioning Index | 12 weeks
  Assesses sexual concerns (e.g., arousal, desire, satisfaction) over the past month
The Greene Climacteric Scale - Sexual Concerns | 12 weeks
  The GCS includes an item that assesses sexual concerns in the past week
The Utian Quality of Life Scale | 12 weeks
  Quality of life will be assessed through The Utian Quality of Life Scale (Utian et al, 2002) is a self-report questionnaire which contains four domains namely, occupational, health, emotional, and sexual in addition to a total score representing quality of life. The current study aims to explore whether CBGT for menopausal symptoms significantly improves quality of life compared to pre-treatment and wait list controls.
Dysfunctional Attitudes Scale (DAS) | 12 weeks
  The Dysfunctional Attitudes Scale (DAS; Weissman, 1979) will be used to assess common beliefs about the self, others, and the future that are considered risk factors of depressive symptoms.
Depression Anxiety Stress Scale (DASS) | 12 weeks
  The Depression Anxiety Stress Scale (DASS; Lovibond & Lovibond, 1995) is a self-report questionnaire that assesses three negative emotional states using three scales (depression scale, anxiety scale, and stress scale). The DASS will be used to explore whether CBGT for menopausal symptoms significantly reduces depressive, anxious, and stress related symptoms, as captured by the DASS, compared to pre-treatment and wait-list controls.
Clinical Global Impression Scale (CGI) | 12 weeks
  Global severity of illness and change in clinical condition will be assessed using the Clinical Global Impression Scale (CGI; Guy, 1976). The current study aims to explore whether CBGT for menopausal symptoms significantly improves global illness severity, as captured by the CGI, compared to pre-treatment and wait-list controls.
Beck Anxiety Inventory (BAI) | 12 weeks
  Changes in subjective somatic or panic-related symptoms of anxiety will be assessed using the Beck Anxiety Inventory (BAI; Beck, 1993). The current study aims to explore whether CBGT for menopausal symptoms significantly reduces anxiety symptoms, as captured by the BAI, compared to pre-treatment and wait-list controls.
Hot Flash Rating Scale: Frequency & Problem Rating Scale (HFRS-FP) | 12 weeks
  Changes in frequency of and distress related to hot flashes will be assessed using the Hot Flash Rating Scale: Frequency & Problem Rating Scale (HFRS-FP; Hunter & Liao, 1995). The current study aims to explore whether CBGT for menopausal symptoms reduces the frequency and distress of hot flashes, as captured by the HFRS-FP, compared to pre-treatment and wait-list controls.
Hot Flash Behaviour Scale (HFBehS) | 12 weeks
  Changes in behavioural reactions to menopausal hot flashes and night sweats will be assessed using the Hot Flash Behaviour Scale (HFBehS; Hunter & Ayers, 2011). The current study aims to explore whether CBGT for menopausal symptoms has an impact on behavioural reactions to menopausal vasomotor symptoms (hot flashes/ night sweats), as captured by the HFBehS, compared to pre-treatment and wait-list controls.
Born Steiner Irritability Scale | 12 weeks
  The Born Steiner Irritability Scale (Born et al., 2004) is a female specific, self-report measure that will be used to assess changes in irritability (annoyance, anger, tension, hostility, and sensitivity to noise and touch). The current study aims to examine whether CBGT for menopausal symptoms is effective in significantly reducing irritability as captured by the Born Steiner Irritability scale, compared to pre-treatment and wait-list controls.
Menopause Representation Questionnaire (MRQ) | 12 weeks
  Cognitions about menopause including those about identity, consequences, time frame and perceptions of control and cure will be assessed using the Menopause Representation Questionnaire (MRQ; Hunter & Dea, 2010). The current study aims to explore whether CBGT for menopausal symptoms has an impact on cognitions about menopause, as captured by the MRQ, compared to pre-treatment and wait-list controls.
Hot Flash Belief Scale (HFBS) | 12 weeks
  Thoughts associated with the menopausal experience of hot flushes and night sweats will be assessed using the Hot Flash Belief Scale (HFBS; Rendall et al. 2008). The current study aims to explore whether CBGT for menopausal symptoms has an impact on beliefs and thoughts associated with hot flushes and night sweats, as captured by the HFBS, compared to pre-treatment and wait-list controls.
Anxiety Sensitivity Index-3 (ASI-3) | 12 weeks
  Changes in anxiety sensitivity will be measured using the Anxiety Sensitivity Index-3 (ASI-3; Taylor et al., 2007). The current study aims to explore whether CBGT for menopausal symptoms significantly reduces fear of anxiety-related situation, as captured by the ASI-3, compared to pre-treatment and wait-list controls.
Couples Satisfaction Index (CSI-32) | 12 weeks
  Changes in relationship satisfaction will be assessed using the Couples Satisfaction Index (CSI-32; Funk & Rogge, 2007). The current study aims to explore whether CBGT for menopausal symptoms improves relationship satisfaction, as captured by the CSI-32, compared to pre-treatment and wait-list controls.
Client Satisfaction Questionnaire (CSQ) | 12 weeks
  Participant satisfaction with the CGBT for menopausal symptoms treatment will be assessed using the Client Satisfaction Questionnaire (CSQ; Larsen et al., 1979).

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Green, PhD, C.Psych, Principal Investigator — St. Joseph's Health Care
Locations (1):
- Women's Health Concerns, St. Joseph's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Donegan E, Frey BN, McCabe RE, Streiner DL, Fedorkow DM, Furtado M, Green SM. Impact of the CBT-Meno protocol on menopause-specific beliefs, dysfunctional attitudes, and coping behaviors. Menopause. 2022 Aug 1;29(8):963-972. doi: 10.1097/GME.0000000000002003. PMID 35881942
- [Derived] Green SM, Donegan E, McCabe RE, Fedorkow DM, Streiner DL, Frey BN. Objective and subjective vasomotor symptom outcomes in the CBT-Meno randomized controlled trial. Climacteric. 2020 Oct;23(5):482-488. doi: 10.1080/13697137.2020.1737929. Epub 2020 Apr 17. PMID 32299247